CLINICAL TRIAL: NCT00258752
Title: Prevention of Depression in Adolescents
Brief Title: Comparison of Three Therapy-Based Interventions for Preventing Depression in Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Rutgers University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: K23MH071320 (NIH); K23MH071320 (NIH); DSIR 8K-RTCT
Record Dates: First submitted 2005-11-23; First posted 2005-11-28 (Estimated); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Depression
Keywords: Prevention; Adolescent
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Interpersonal Psychotherapy-Adolescent Skills Training (IPT-AST)
  Interventions: Behavioral: IPT-AST
- 2 (Experimental): Enhanced IPT-AST
  Interventions: Other: Enhanced IPT-AST
- 3 (Active Comparator): Typical school counseling
  Interventions: Other: School counseling

INTERVENTIONS:
Behavioral: IPT-AST — IPT-AST is a school based group treatment program that focuses on prevention, psychoeducation, and interpersonal skill building.
  Arms: 1
Other: Enhanced IPT-AST — Enhanced IPT-AST entails IPT-AST plus three parent-adolescent sessions.
  Arms: 2
Other: School counseling — Usual care consists of standard treatments, including individual counseling with guidance counselor.
  Arms: 3

SUMMARY:
This study will compare Interpersonal Psychotherapy-Adolescent Skills Training (IPT-AST), IPT-AST plus parent involvement (Enhanced IPT-AST), and Usual Care for the prevention of adolescent depression.

DETAILED DESCRIPTION:
Depression is a serious medical illness that is difficult to diagnose and treat, especially in children and adolescents. Signs of depression in children may include the following behaviors: pretending to be sick; refusing to go to school; clinging to a parent; or worrying that a parent may die. Older children may sulk, behave inappropriately at school, act in a negative or grouchy manner, or feel misunderstood. Because normal behaviors vary from one childhood stage to another, it can be difficult to determine whether a child is going through a temporary "phase" or is suffering from depression. This study will compare IPT-AST, Enhanced IPT-AST, and Usual Care for the prevention of adolescent depression.

Participation in this single-blind study will last approximately 21 months. Participants will be randomly assigned to receive either IPT-AST, Enhanced IPT-AST, or Usual Care for 12 weeks. IPT-AST is a school-based group intervention program that focuses on prevention, psychoeducation, and interpersonal skill-building. Enhanced IPT-AST will entail IPT-AST plus three parent-adolescent sessions. Usual Care will consist of standard treatments and will not include IPT-AST. Study visits will occur before and during the intervention at baseline and Weeks 6 and 12. Follow-up visits will occur 6, 12, and 18 months post-intervention. Study visit assessments will include depression symptoms, anxiety symptoms, psychiatric diagnoses, overall functioning, social adjustment, parent-child conflict, perceived support from parents and peers, and service utilization.

ELIGIBILITY:
Inclusion Criteria:

* Between grades 7 and 10 in school
* Score of at least 16 on the Center for Epidemiologic Studies Short Depression Scale (CES-D)
* Currently experiencing at least 2 symptoms on the K-SADS depression section, one of which is either depressed mood, irritability, or an inability to feel pleasure during normal activities
* Score of at least 61 on the Children's Global Assessment Scale (CGAS), indicating mild to moderate impairment
* English-speaking

Exclusion Criteria:

* Score of 15 or less on the CES-D scale
* Currently experiencing fewer than 2 depression symptoms on the K-SADS or 2 or more symptoms on the K-SADS with no report of depressed mood, irritability, or anhedonia
* Attempted suicide or self-mutilation in the year prior to study entry
* Current active suicidal ideation and/or history of a clinically significant suicidal behavior (i.e., with intent to die and high medical lethality) or repeated patterns of self-injurious behavior
* Current major depressive disorder or dysthymia as determined by K-SADS
* Current DSM-IV diagnosis of psychosis, substance abuse or dependence, bipolar disorder, obsessive compulsive disorder, post-traumatic stress disorder, panic disorder, or conduct disorder as determined by K-SADS
* Score of 60 or less on the CGAS, indicating substantial functional impairment

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 57 (Actual)
Dates: Start 2005-11; Primary Completion 2008-01 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Score on the Center for Epidemiologic Studies Depression Scale | Measured immediately post-treatment and at Months 6, 12, and 18 follow-ups
Rating on Children's Global Assessment Scale | Measured immediately post-treatment and at Months 6, 12, and 18 follow-ups
Depression diagnoses on the Kiddie Schedule for Affective Disorders and Schizophrenia (K-SADS) diagnostic instrument | Measured immediately post-treatment and at Months 6, 12, and 18 follow-ups

SECONDARY OUTCOMES:
Score on the Conflict Behavior Questionnaire | Measured immediately post-treatment and at Months 6, 12, and 18 follow-ups
Score on the Social Adjustment Scale | Measured immediately post-treatment and at Months 6, 12, and 18 follow-ups
Score on the Perceived Social Support scale | Measured immediately post-treatment and at Months 6, 12, and 18 follow-ups

CONTACTS AND LOCATIONS:
Overall Officials: Jami F. Young, PhD, Principal Investigator — Rutgers University
Locations (2):
- United States (2):
  - Rutgers University, Piscataway, New Jersey
  - New York State Psychiatric Institute, New York, New York